CLINICAL TRIAL: NCT04186598
Title: Multicenter Randomized Double-Blind Control Trial Evaluating the Utility of Continuous Positive Airway Pressure (CPAP) in the Treatment of High Altitude Pulmonary Edema (HAPE)
Brief Title: Evaluating the Utility of Continuous Positive Airway Pressure in the Treatment of High Altitude Pulmonary Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CommonSpirit Health (Other)
Collaborators: Pulmodyne, Inc. (Unknown)
Responsible Party: Principal Investigator, Todd Bolotin, Principal Investigator, CommonSpirit Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1389613
Record Dates: First submitted 2019-12-01; First posted 2019-12-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Continuous Positive Airway Pressure; High Altitude Pulmonary Edema
MeSH Terms: conditions — Altitude Sickness | interventions — Nifedipine; Positive-Pressure Respiration

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Standard CPAP systems and control CPAP systems that provide high flow oxygen without PEEP
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental: CPAP (Experimental): Participants will be treated with CPAP. All patients will be treated with nifedipine unless there is a contraindication like hypotension and bradycardia.
  Interventions: Device: CPAP mask system; Drug: Nifedipine 30 MG
- Control: High flow oxygen (Placebo Comparator): Participants will be treated with an altered CPAP mask that will deliver high flow oxygen. All patients will be treated with nifedipine unless there is a contraindication like hypotension and bradycardia.
  Interventions: Drug: Nifedipine 30 MG; Device: CPAP mask system without PEEP

INTERVENTIONS:
Device: CPAP mask system — Intervention group will receive 15cm of H2O of positive end expiratory pressure
  Arms: Experimental: CPAP
Drug: Nifedipine 30 MG — All participants will receive this intervention
Device: CPAP mask system without PEEP — Placebo group will receive high flow oxygen via altered CPAP mask system without providing any positive end expiratory pressure
  Arms: Control: High flow oxygen

SUMMARY:
The primary objective is to evaluate the efficacy of continuous positive pressure on resolution of high-altitude pulmonary edema vs high flow oxygen. The secondary objective is to derive an incidence of high-altitude pulmonary edema based on the elevation and timing from which the subject arrives. Additionally, in a convenience sample of the base study population, an ultrasound evaluation for the presence of B lines in the lungs will be conducted after 2 hours.

DETAILED DESCRIPTION:
Multicenter, double-blinded, randomized control trial. Enrollment is based on presentation to one of the treating facilities with clinical signs and symptoms of high-altitude pulmonary edema with a recent arrival at high altitude, an oxygen saturation below 85%, and radiographic evidence of noncardiogenic pulmonary edema. A total of 264 patients will be randomized 1:1 across 2 study arms: a CPAP mask set to 15cm H2O and an altered CPAP mask in which the pressure valve has been modified to deliver no positive pressure. All patients will be treated with 30mg nifedipine XR. Except for the application of positive pressure, all other interventions are performed in the context of everyday clinical practice, and thus will be equivalent for participants in both arms. Patients will be evaluated every 30 minutes for their ability to maintain an oxygen saturation of 92% with a normal respiratory rate and no signs of increased work of breathing on 2 liters of nasal cannula oxygen for a total of up to a maximum treatment length of 2 hours. The primary efficacy endpoint will be assessed every 30 minutes for 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or greater
* Oxygen saturation below 85%
* Recent arrival to high altitude
* Dyspnea and cough
* Xray revealing non-cardiogenic pulmonary edema

Exclusion Criteria:

* Pregnancy
* Age below 18
* Patients with respiratory failure requiring intubation
* Patients with altered mental status
* Patients with impaired decision-making capacity
* Patients with a history of congestive heart failure, CAD, COPD, asthma, known current pneumonia
* Extreme facial hair precluding application of CPAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Time to resolution of HAPE | 2 hours
  The amount of time it took to maintain oxygen saturation over 92% on 2L NC oxygen

SECONDARY OUTCOMES:
Presence or absence of ultrasound detectable B lines | 2 hours
  A convenience sample of the total study population will have a bedside pulmonary ultrasound at time zero and two hours
Characterization of time at altitude to development of HAPE | 2 hours
  A descriptive measurement of the time since the patient arrived at altitude until the development of HAPE
Incidence of HAPE by native altitude and reported sleeping altitude | 2 hours
  Data will be collected and analyzed to seek a relationship between the subjects home altitude and the altitude of their sleep while at high altitude

CONTACTS AND LOCATIONS:
Overall Officials: Todd Bolotin, MD, Principal Investigator — CommonSpirit Health
Locations (1):
- Breckenridge Medical Center, Breckenridge, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Murdoch DR. Prevention and Treatment of High-altitude Illness in Travelers. Curr Infect Dis Rep. 2004 Feb;6(1):43-49. doi: 10.1007/s11908-004-0023-4. PMID 14733848
- [Background] Gonzalez Garay A, Molano Franco D, Nieto Estrada VH, Marti-Carvajal AJ, Arevalo-Rodriguez I. Interventions for preventing high altitude illness: Part 2. Less commonly-used drugs. Cochrane Database Syst Rev. 2018 Mar 12;3(3):CD012983. doi: 10.1002/14651858.CD012983. PMID 29529715
- [Background] Basnyat B, Murdoch DR. High-altitude illness. Lancet. 2003 Jun 7;361(9373):1967-74. doi: 10.1016/S0140-6736(03)13591-X. PMID 12801752
- [Background] Gallagher SA, Hackett PH. High-altitude illness. Emerg Med Clin North Am. 2004 May;22(2):329-55, viii. doi: 10.1016/j.emc.2004.02.001. PMID 15163571
- [Background] Nieto Estrada VH, Molano Franco D, Medina RD, Gonzalez Garay AG, Marti-Carvajal AJ, Arevalo-Rodriguez I. Interventions for preventing high altitude illness: Part 1. Commonly-used classes of drugs. Cochrane Database Syst Rev. 2017 Jun 27;6(6):CD009761. doi: 10.1002/14651858.CD009761.pub2. PMID 28653390
- [Background] Stoltzfus S. The role of noninvasive ventilation: CPAP and BiPAP in the treatment of congestive heart failure. Dimens Crit Care Nurs. 2006 Mar-Apr;25(2):66-70. doi: 10.1097/00003465-200603000-00006. PMID 16552275
- [Background] Luks AM, Auerbach PS, Freer L, Grissom CK, Keyes LE, McIntosh SE, Rodway GW, Schoene RB, Zafren K, Hackett PH. Wilderness Medical Society Clinical Practice Guidelines for the Prevention and Treatment of Acute Altitude Illness: 2019 Update. Wilderness Environ Med. 2019 Dec;30(4S):S3-S18. doi: 10.1016/j.wem.2019.04.006. Epub 2019 Jun 24. PMID 31248818
- [Background] Johnson PL, Johnson CC, Poudyal P, Regmi N, Walmsley MA, Basnyat B. Continuous positive airway pressure treatment for acute mountain sickness at 4240 m in the Nepal Himalaya. High Alt Med Biol. 2013 Sep;14(3):230-3. doi: 10.1089/ham.2013.1015. PMID 24067184
- [Background] Hebert PC, Stanbrook M. Indication creep: physician beware. CMAJ. 2007 Sep 25;177(7):697, 699. doi: 10.1503/cmaj.071223. Epub 2007 Sep 5. No abstract available. PMID 17823137
- [Background] Walmsley M. Continuous positive airway pressure as adjunct treatment of acute altitude illness. High Alt Med Biol. 2013 Dec;14(4):405-7. doi: 10.1089/ham.2013.1059. PMID 24377348
- [Derived] Bolotin T, Subedi S, Dahal S, Walker C, Chung K, Martz A, Gemmel D, Chopra Q, Donley C. High Altitude Pulmonary Edema Response to Continuous Airway Positive Pressure: A Randomized Controlled Trial: The HAPER CAPER Trial. Acad Emerg Med. 2025 Nov;32(11):1215-1223. doi: 10.1111/acem.70126. Epub 2025 Sep 12. PMID 40938265